CLINICAL TRIAL: NCT04739839
Title: Risk Factors for Low Back Pain in Adults a 23-year Prospective Cohort Study of 14-15-year-old Schoolchildren.
Status: Terminated | Type: Observational
Why Stopped: Lack of responders
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Marius Henriksen, Clinical professor, Frederiksberg University Hospital
Other Study IDs: Western Zealand Cohort
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2022-01

CONDITIONS: Low Back Pain
Keywords: low back pain; prevalence; illness perception; quality of life; cohort study; survey
MeSH Terms: conditions — Low Back Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Inception cohort, former pupils in different schools in Western Zealand: 1327 former Western Zealand pupils (originally 1389). Aged 14-15 in 1997. This is the first follow up on this cohort.
  Interventions: Other: survey questionnaire

INTERVENTIONS:
Other: survey questionnaire — Questionnaire focusing on low back pain in relation to life style, physical activity level, illness perception and quality of life.

SUMMARY:
The incidence of low back pain (LBP) is increasing and prognostic factors for developing LBP are unclear. Based on questionnaires, different prognostic factors are being explored over time.

DETAILED DESCRIPTION:
Despite the massive efforts of trying to find predictors and prevention for LBP, it remains to be clarified, why some individuals develop severely disabling low back pain while others never experience noteworthy back pain.

There is no evidence that numbers of chronically affected individuals have diminished; rather, the incidence of LBP has increased continuously over the last 20 years, which is also reflected in rising numbers of lumbar surgical treatments and rising costs due to health care expenses and sick leave. Hence, prevention of LBP in the working population seems more urgent than ever.

As LBP is undoubtedly a multifaceted disorder that tends to fluctuate throughout life, there is a need for longitudinal research, exploring the effect of both lifestyle and psychosocial factors on the development of chronic low back pain.

The main aims of this study is to identify the prevalence of low back pain and identify whether a history of low back pain during adolescence represents an increased risk of experiencing low back pain later in life.

ELIGIBILITY:
Inclusion Criteria:

* Being a member of the original Western Zealand cohort
* Ability to understand and write in Danish
* Having access to the Danish digital mail system "e-Boks". (Access to e-Boks is mandatory in Denmark unless you have special needs)

Exclusion Criteria:

We have no formal exclusion criterias

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is an inception cohort where all participants will be around 38 years
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence of low back pain | Measured once at study baseline
  Amount of respondents reporting low back pain within last month

SECONDARY OUTCOMES:
Incidence of severe low back pain | Measured once at study baseline
  Amount of respondents reporting low back pain more than thirty days within last year
Actual low back pain | Measured once at study baseline
  Current low back pain, defined as "the level of pain in your lower back today"
The Brief Illness Perception Questionnaire | Measured once at study baseline
  We use the Danish version of The Brief illness perception questionnaire (B-IPQ). B-IPQ is a generic 9-item questionnaire developed to rapidly assess the cognitive and emotional representations in a variety of illnesses. The first 8 items are scored on a 1-10 numeric rating scale with descriptors (none or extreme) at either end. B-IPQ assesses perceptions on the following five dimensions: Identity, Cause, Timeline, Consequences and Cure-Control. Five of the items assess cognitive illness representations: consequences, timeline, personal control, treatment control, and identity. Two of the items assess emotional representations: concern and emotions. One item assesses illness comprehensibility. Item 9 is a free text field in which the respondent can formulate their beliefs about their condition (cause). We will not use this field in our study. In all questions we replace the word "illness" with "low back pain".
  In this study we explore each B-IPQ item score and not an overall score.
Roland Morris Questionnaire | Measured once at study baseline
  The Roland Morris Questionnaire (RMQ) is designed to assess self-rated physical disability caused by low back pain. It is most sensitive for patients with mild to moderate disability due to acute, sub-acute or chronic low back pain. It is easy to administer and correlates well with other physical disability measures. We used the Danish version (RMQ-Patrick). It has 23 questions with yes/no options and is translated in 2003. A clinically meaningful change on the RMQ ranges from a 2.5- to a 5.0-point improvement (reduction) from baseline has been suggested.
Health related quality of life EQ-5D | Measured once at study baseline
  To assess health related quality of life we apply the Danish version of the EuroQoL 5 dimensions (EQ-5D) questionnaire. EQ-5D is a standardised measure of health status that provides a simple, generic measure of health. It is applicable to a wide range of health conditions and is ideally suited for use in surveys. The EQ-5D consists of a descriptive system comprising 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Standardized answer options are given (3 Likert boxes) and each question is assigned a score from 1 to 3. From the responses an EQ-5D index is calculated. Further a EQ visual analogue scale (EQ VAS) is used to record the respondent's self-rated health on a 0-100 vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine' used as a quantitative measure of health as judged by the individual respondents.
Health related quality of life EQ-5D VAS | Measured once at study baseline
  A visual analogue scale (EQ VAS) is used to record the respondent's self-rated health on a 0-100 vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine' used as a quantitative measure of health as judged by the individual respondents.
Use of CAMs for low back pain | Measured once at study baseline
  Amount of respondents reporting regular use of complementary or alternative treatments (CAMs) for low back pain
Use of exercise for low back pain | Measured once at study baseline
  Amount of respondents doing regular exercise for low back pain
Use of recommended non-pharmacological treatments for low back pain | Measured once at study baseline
  Amount of respondents reporting regular use of recommended non-pharmacological treatments for low back pain
Use of recommended pharmacological treatments for low back pain | Measured once at study baseline
  Amount of respondents reporting regular use of recommended pharmacological treatments for low back pain

CONTACTS AND LOCATIONS:
Locations (1):
- Claus Bomhoff, Copenhagen, DK, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will be available through request to study contact person